CLINICAL TRIAL: NCT00985998
Title: Phase 1 Study of Nimotuzumab in Combination With Cisplatin and Docetaxel for Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Nimotuzumab in Combination With Cisplatin and Docetaxel for Patients With Advanced Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no paticipants enrolled
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-NSCLC-T-0902
Record Dates: First submitted 2009-09-27; First posted 2009-09-29 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: nimotuzumab; non-small cell lung cancer; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nimotuzumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nimotuzumab (Experimental)
  Interventions: Drug: Nimotuzumab and chemotherapy

INTERVENTIONS:
Drug: Nimotuzumab and chemotherapy — The chemotherapy treament：docetaxel( 75mg/m2/d,every21days,for4~6cycles) and cisplatin(total dose 75mg/m2 on day 2,3,4,every21days,for4~6cycles).
  the nimotuzumab treatment:3 levels (200mg/w,400mg/w,600mg/w,weekly,for12~18 weeks).
  Other Names: Nimotuzumab

SUMMARY:
Nimotuzumab (hR3) is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Clinical efficacy has been shown in adult with head and neck cancer. The study assessed the safety, and efficacy of the combination of Nimotuzumab administered concomitantly with chemotherapy in patients with advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Altered expression or constitutive activation of the epidermal growth factor receptor (EGFR/HER1/erbB1) commonly occurs in primary NSCLC, and is often a critical factor in progressive growth and resistance to normal mechanisms of cell death. Epidermal growth factor receptor expression in lung cancer has been correlated with tumor aggressiveness. Clinical trials already suggest that EGFR targeted therapy may improve the antitumor activity of chemotherapy for treatment of lung carcinoma. Monoclonal antibodies specific to EGFR can be combined safely and effectively with chemotherapy. Nimotuzumab (hR3) is a humanized monoclonal antibody (mAb) that binds to the EGFR. In preclinical studies the antibody has shown potent antitumor activity. A previous phase II study in children with high grade brain tumors showed activity of Nimotuzumab as a monotherapeutic agent, even in prognostic very unfavourable diffuse, intrinsic pontine glioma. No drug related side effects were reported. Nimotuzumab (hR3) in combination with radiotherapy for treatment of locally advanced squamous cell carcinomas of the head and neck resulted in high rates of antitumor response, and was accompanied by a favourable safety profile.

This is a dose-escalation study of Nimotuzumab. Nimotuzumab in combination with chemotherapy will be administered to the patients with advanced NSCLC. The patients' blood test and liver and renal function tests will be monitored weekly, a physical exam and reassessment of the tumor will be performed and every 6 weeks. When the total result is the CR or PR, the results of the 6th, 12th, 18th and the 22th week should be compared.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pathologically or cytologically documented stage IIIB or IV NSCLC. Disease must be newly diagnosed .
* Presence of at least 1 uni-dimensionally measurable index lesion,with the longest diameter ≥ 20 mm using conventional computer tomography(CT)/magnetic resonance imaging(MRI)scan or ≥ 10 mm using spiral computed tomography scan.
* Age > 18 and < 65, with ECOG performance status 0-1,and Life expectancy of more than 3 months.
* functions of major organs (haemogram, heart, liver, kidney) are basically normal, White blood count ≥3.5 x 109/L with neutrophils ≥1.5 x 109/L, platelet count≥100 x 109/L, and hemoglobin ≥100g/L. Total bilirubin ≤1.5 times upper limit of normal (ULN) range; alkaline phosphatase(ALP)≤ 2.5 times ULN or ≤5 times ULN (liver metastasis); Transaminases AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN or ≤ 5 times ULN (liver metastasis). serum creatinine ≤ 1.2 times ULN, blood urea nitrogen≤ 1.2 times ULN.
* both female and male patients must use adequate methods of contraception.
* without other malignancy history, except curative carcinoma in situ of cervix and skin basal cell carcinoma.
* willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Previous radiotherapy（except the radiotherapy of brain metastasis）, Previous chemotherapy or anticancer biotherapy , Participation other clinical trials within 1 month prior to inclusion in the trial.
* With only unmeasureable lesion, ie, hydrothorax, ascites, lymphangitis carcinomatous, diffuse liver metastasis, bony metastasis; no measureable lesion or the lesion could not be determined.
* Pregnant or breast-feeding women or using a prohibited contraceptive method.
* With Symptomatic brain metastasis not controlled.
* with an uncontrolled seizure disorder, or active centre neurological disease, or Psychiatric disease affected cognitive ability; physiogenic or pathological dystrophinopathies, chronic diarrhea, cachexia.
* with significant history of cardiac disease, i.e., congestive heart failure, angina requiring medication, uncontrolled cardiac ventricular arrythmias, heart valve disease, serious myocardial infarction, uncontrolled hypertension.
* With other serious internal diseases or uncontrolled infection.
* With drug addition,ie,drug-taking,drug-taking for long time;with AIDS.
* With organ transplantation,or using adrenocortical hormone or immunosuppressive agents for long time.
* With history of serious allergic or allergy.
* Not fit for the clinical trial judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity of this new treatment. Both acute and chronic toxicity will be evaluated. | within study period

SECONDARY OUTCOMES:
To determine the complete response rate、partial rate、disease response rate、disease control rate in the patients subject to treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Professor, Principal Investigator — 86-10-87788121
Locations (1):
- Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China